CLINICAL TRIAL: NCT02910882
Title: A Phase II Study Combining PEGPH20 With Concurrent Gemcitabine and Radiotherapy in Patients With Localized, Unresectable Pancreatic Adenocarcinoma
Brief Title: PEGPH20 Plus Gemcitabine With Radiotherapy in Patients With Localized, Unresectable Pancreatic Cancer
Acronym: HALO-IST
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety
Sponsor: Scripps Health (Other)
Responsible Party: Principal Investigator, Darren Sigal, MD, Principal Investigator, Scripps Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEGPH20-GEM-XRT
Record Dates: First submitted 2016-08-12; First posted 2016-09-22 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Pancreatic Adenocarcinoma Non-resectable
Keywords: Pancreas Cancer; Unresectable; Chemoradiation; PEGPH20
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — PEGPH20; Gemcitabine; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Cohort I (PEGPH20 Dose Escalation + Gemcitabine and Concurrent Radiotherapy), First 3 Patients:
  An abbreviated sequential dose escalation schema for the first 3 patients (each subsequent patient will be accrued only after no dose limiting toxicities are found in the first 2 weeks of concurrent therapy for the previous patient).
  Intravenous (IV) PEGPH20, per dose escalation guidelines for first 3 patients; Intravenous (IV) Gemcitabine (Standard Regimen); Radiotherapy (Standard Regimen);
  Cohort II (PEGPH20 + Gemcitabine and Concurrent Radiotherapy), Patients 4 - 10:
  IV PEGPH20, per dosing level determined in dose escalation (Cohort I); IV Gemcitabine (Standard Regimen); Radiotherapy (Standard Regimen);
  Interventions: Drug: PEGylated Recombinant Human Hyaluronidase (PEGPH20); Drug: Gemcitabine; Radiation: Radiation

INTERVENTIONS:
Drug: PEGylated Recombinant Human Hyaluronidase (PEGPH20) — PEGPH20 Dosing (Cohort I, Dose Escalation, First 3 patients): Administered as an IV infusion over 10 minutes (+/- 2 Minutes), approximately 1mL/minute:
  Dose level 1 - 1 mcg/kg; Dose level 2 - 1.6 mcg/kg; Dose level 3 - 3 mcg/kg.
  PEGPH20 Dosing (Cohort II, Patients 4-10): Administered at a dose of 3 mcg/kg as an IV infusion over 10 minutes (+/- 2 Minutes), approximately 1mL/minute.
  Dosing Schedule: Twice per week beginning Day #1 for 8 doses, then weekly until end of radiotherapy.
  Other Names: PEGylated rHuPH20
Drug: Gemcitabine — Gemcitabine Dosing: Administered at a dose of 600 mg/m2 as an IV infusion over 30 - 60 minutes with standard antiemetic pre-medication. If administered on PEGPH20 day, Gemcitabine will be infused 2-4 Hours after PEGPH20 infusion is completed.
  Dosing Schedule: Weekly, beginning Day #2, per standard regimen.
  Other Names: Gemzar
Radiation: Radiation — Radiotherapy, beginning Day #2, delivered at 1.8 Gy per fraction, 5 fractions per week (Monday - Friday), until a total dose of 50.4 to 54 Gy for up to 6 Weeks.

SUMMARY:
This is a single arm phase II trial assessing the potential activity of combination PEGPH20 plus Gemcitabine with radiotherapy in ten patients with localized, unresectable pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
This is a pilot trial evaluating the safety and potential efficacy of PEGylated Recombinant Human Hyaluronidase (PEGPH20) plus concurrent Gemcitabine and radiotherapy. Recognizing that PEGPH20 has not been previously delivered with radiotherapy but is unlikely to contribute to increased toxicities, this trial will have an abbreviated sequential dose escalation schema for the first three patients. PEGPH20 will be given twice per week for the first 28 days and then weekly for another 2 weeks during radiotherapy. Gemcitabine will be delivered weekly at the first day of radiotherapy and continued weekly, per published literature. Patients will remain on study for three months. The duration of active treatment with PEGPH20 and Gemcitabine plus radiotherapy will continue for 5-6 weeks. Efficacy outcome will occur 6-8 weeks after the completion of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy all the following inclusion criteria to be enrolled in the study:

1. Signed, written Institutional Review Board/Ethics Committee-approved Informed Consent Form;
2. For men and women of reproductive potential, agreement to use an effective contraceptive method from the time of screening and throughout their time on study. Effective contraceptive methods consist of prior sterilization, intra-uterine device, oral or injectable contraceptives, and/or barrier methods. Abstinence alone is not considered an adequate contraceptive measure for the purposes of this study;
3. Patients with previously untreated localized, unresectable histologically confirmed pancreatic adenocarcinoma (unresectable will be defined as locally advanced disease or when patients cannot have or refuse surgery);
4. Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L;
5. Platelets ≥ 100 x 109/L;
6. Hgb ≥ 9 g/dL;
7. Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5 x [Upper Limit of Normal (ULN)];
8. Bilirubin ≤ 1.5 x ULN;
9. GFR ≥ 30 mL/min;
10. Patient has no clinically significant abnormalities in urinalysis results;
11. Patient has acceptable coagulation status as indicated by a Prothrombin Time (PT) and Partial Thromboplastin Time (PTT) within 15% of normal limits;
12. Eastern Cooperative Oncology Group (ECOG) ≤ 2

Exclusion Criteria:

Subjects are ineligible for enrollment if they meet any of the following exclusion criteria:

1. Clinical evidence of deep vein thrombosis (DVT), pulmonary embolism (PE) or other known thromboembolic (TE) event present during the screening period;
2. Any prior history of cerebrovascular accident, transient ischemic attack, or pre-existing carotid artery disease.
3. Known allergy to hyaluronidase;
4. Current use of megestrol acetate (use within 10 days of Day 1);
5. Contraindication to heparin including prior heparin induced thrombocytopenia (HIT), recent CNS bleed; intracranial or spinal lesion at high risk for bleeding; severe platelet dysfunction; recent major operation at high risk for bleeding; underlying hemorrhagic coagulopathy; high risk for falls; potential need for spinal anesthesia/lumbar puncture; active bleeding;
6. Women currently pregnant or breastfeeding;
7. Intolerance to dexamethasone;
8. Inability to comply with study and follow-up procedures as judged by the Investigator;
9. Patient has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy;
10. Patient has known infection with HIV, hepatitis B, or hepatitis C;
11. Patient has a history of allergy or hypersensitivity to any of the agents they are supposed to receive (or to any of the excipients for those agents);
12. Patient has serious medical risk factors involving any of the major organ systems such that the investigator considers it unsafe for the patient to receive an experimental research drug, these can include New York Heart Association Functional Class ≥ 3, myocardial infarction within the past 12 months before screening, pre-existing atrial fibrillation, symptomatic COPD.
13. Patient is unwilling or unable to comply with study procedures.

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Related Adverse Events (AEs) | Up to 8 Weeks After the End of Treatment
  Adverse events will be assessed weekly, from Day1 Treatment through up to 8 weeks after the end of treatment. Safety will be assessed during the study by evaluation of AEs, clinical safety laboratory tests (hematology, blood chemistry (including C-reactive protein [CRP]), coagulation, urinalysis, and PEGPH20 immunogenicity), vital signs, 12-lead ECGs, and physical examinations.
  The severity of AEs will be graded by Investigators using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03

SECONDARY OUTCOMES:
Overall Tumor Response Rate | Change from Baseline through 8 Weeks After End of Radiation Therapy
  CT Chest/Abdomen/Pelvis will be completed at End of Study Visit. End of Study visit will be done 6-8 weeks after the last day of radiotherapy. The evaluation of overall lesion response will be a composite of the target lesion response, non-target lesion response and presence of new lesions, per RECIST 1.1 criteria.
Conversion to Resectability Rate | Up to 8 Weeks After End of Radiation Therapy
  Number of enrolled subjects completing at least 2 weeks of PEGPH20 plus concurrent gemcitabine and radiotherapy who meet institutional surgical criteria for surgical resectability, as determined by End of Study CT imaging. End of Study CT imaging will be done up to 8 weeks after the end of radiation therapy.
Carcinoembryonic Antigen (CEA) Response | Change from Day 1 through 8 Weeks After End of Treatment
  Change in CEA serum levels from Day 1 through 8 weeks after end of treatment will be assessed.
CA 19-9 Response | Change from Day 1 through 8 Weeks After End of Treatment
  Change in CA 19-9 serum levels from Day 1 through 8 weeks after end of treatment will be assessed.
Determine the Maximum or Peak Plasma PEGPH20 Concentration (cmax) at End of Infusion | At Specific Timepoints from Day 1 through Day 39 During Treatment
  Maximum Plasma PEGPH20 concentration (cmax) will be analyzed in all patients, at the following time points:
  Day 1: Pre-Dose; Day 1 Post-Dose @ 1hr, 2hr, 6hr; Day 2 (24Hr Post Dose); Day 3 (48Hr Post Dose); Day 4 (72Hr Post Dose); Day 8: Pre-Dose; Day 9 (24Hr Post Dose); Day 10 (48Hr Post Dose); Day 11 (72 Hr Post Dose); Day 36: Pre-Dose; Day 37 (24 Hr Post Dose); Day 38 (48Hr Post Dose); Day 39 (72 Hr Post Dose);
  Pharmacokinetic (PK) data will analyzed by non-compartmental analysis (NCA).
Determine Plasma PEGPH20 Area Under the Curve (AUC) After Day 1 PEGPH20 Infusion | At Specific Timepoints from Day 1 through Day 39 During Treatment
  Plasma PEGPH20 Area Under the Curve (AUC) will be analyzed in all patients, at the following time points:
  Day 1: Pre-Dose; Day 1 Post-Dose @ 1hr, 2hr, 6hr; Day 2 (24Hr Post Dose); Day 3 (48Hr Post Dose); Day 4 (72Hr Post Dose); Day 8: Pre-Dose; Day 9 (24Hr Post Dose); Day 10 (48Hr Post Dose); Day 11 (72 Hr Post Dose); Day 36: Pre-Dose; Day 37 (24 Hr Post Dose); Day 38 (48Hr Post Dose); Day 39 (72 Hr Post Dose);
  Pharmacokinetic (PK) data will analyzed by non-compartmental analysis (NCA).
Determine the Maximum or Peak Plasma Hyaluronan Concentration (cmax) After First Dose of PEGPH20 | At Specific Timepoints from Day 1 through Day 39 During Treatment
  Plasma Hyaluronan (HA) will be analyzed in all patients, at the following time points:
  Day 1: Pre-Dose; Day 2 (24Hr Post Dose); Day 3 (48Hr Post Dose); Day 4 (72Hr Post Dose); Day 8: Pre-Dose; Day 9 (24Hr Post Dose); Day 10 (48Hr Post Dose); Day 11 (72 Hr Post Dose); Day 36: Pre-Dose; Day 37(24 Hr Post Dose); Day 38(48Hr Post Dose); Day 39 (72 Hr Post Dose);
  Hyaluronan pharmacodynamic (PD) data will analyzed by non-compartmental analysis (NCA).
Determine Plasma Hyaluronan Area Under Effect Curve (AUEC) After First Dose of PEGPH20 | At Specific Timepoints from Day 1 through Day 39 During Treatment
  Plasma Hyaluronan (HA) will be analyzed in all patients, at the following time points:
  Day 1: Pre-Dose; Day 2 (24Hr Post Dose); Day 3 (48Hr Post Dose); Day 4 (72Hr Post Dose); Day 8: Pre-Dose; Day 9 (24Hr Post Dose); Day 10 (48Hr Post Dose); Day 11 (72 Hr Post Dose); Day 36: Pre-Dose; Day 37(24 Hr Post Dose); Day 38(48Hr Post Dose); Day 39 (72 Hr Post Dose);
  Hyaluronan pharmacodynamic (PD) data will analyzed by non-compartmental analysis (NCA).

CONTACTS AND LOCATIONS:
Overall Officials: Darren S Sigal, MD, Principal Investigator — Scripps Health/Scripps Clinic
Locations (1):
- Scripps Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baumgartner G, Gomar-Hoss C, Sakr L, Ulsperger E, Wogritsch C. The impact of extracellular matrix on the chemoresistance of solid tumors--experimental and clinical results of hyaluronidase as additive to cytostatic chemotherapy. Cancer Lett. 1998 Sep 11;131(1):85-99. PMID 9839623
- [Background] Hingorani S, Harris WP, Beck JT, Berdov BA, Wagner SA, Pshevlotskyet EM, et al. Final Results of a Phase 1b Study of Gemcitabine Plus PEGPH20 in Patients With Stage IV Previously Untreated Pancreatic Cancer. ASCO 2015 Gastrointestinal Cancers Symposium, Poster Abstract 359.
- [Background] Loehrer PJ Sr, Feng Y, Cardenes H, Wagner L, Brell JM, Cella D, Flynn P, Ramanathan RK, Crane CH, Alberts SR, Benson AB 3rd. Gemcitabine alone versus gemcitabine plus radiotherapy in patients with locally advanced pancreatic cancer: an Eastern Cooperative Oncology Group trial. J Clin Oncol. 2011 Nov 1;29(31):4105-12. doi: 10.1200/JCO.2011.34.8904. Epub 2011 Oct 3. PMID 21969502
- [Background] Vaupel P, Thews O, Hoeckel M. Treatment resistance of solid tumors: role of hypoxia and anemia. Med Oncol. 2001;18(4):243-59. doi: 10.1385/MO:18:4:243. PMID 11918451
- [Background] Provenzano PP, Hingorani SR. Hyaluronan, fluid pressure, and stromal resistance in pancreas cancer. Br J Cancer. 2013 Jan 15;108(1):1-8. doi: 10.1038/bjc.2012.569. Epub 2013 Jan 8. PMID 23299539
- [Background] Li X, Jiang P, Symons R, et al. Pegylated human recombinant hyaluronidase PH20 reduces solid tumor hypoxia [abstract]. Cancer Res 2012; 72(8 Suppl): Abstract 3796.
- [Background] Li X. PEGylated human recombinant hyaluronidase (PEGPH20) removes peritumoral hyaluronan and increases the efficacy of chemotherapy and radiotherapy in an experimental brain metastasis model [abstract]. Cancer Res 2009; 69 (9 Suppl): Abstract 262.